CLINICAL TRIAL: NCT00247273
Title: A Phase III, Multicenter, Double-blind, Randomized, Active-controlled, Parallel Group, Non-inferiority Study Comparing 150 mg Risedronate Monthly With 5 mg Risedronate Daily in the Treatment of Postmenopausal Osteoporosis (PMO)
Brief Title: A Study of Monthly Risedronate for Osteoporosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Warner Chilcott (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2005032; EFC6062 AND HMRF004M/3001
Record Dates: First submitted 2005-10-28; First posted 2005-11-01 (Estimated); Results first posted 2011-06-21 (Estimated); Last update posted 2013-04-22 (Estimated); Status verified 2013-04

CONDITIONS: Postmenopausal Osteoporosis
Keywords: randomized controlled trial, osteoporosis, risedronate
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporosis | interventions — Risedronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): 5 mg risedronate, once daily for 2 years
  Interventions: Drug: risedronate
- 2 (Experimental): 150 mg risedronate taken once a month for 2 years
  Interventions: Drug: risedronate

INTERVENTIONS:
Drug: risedronate — tablet, 5 mg risedronate, once a day for 2 years
  Arms: 1
Drug: risedronate — oral, 150 mg risedronate, once a month for 2 years

SUMMARY:
The purpose of this trial is to study the efficacy of a single-dose monthly dosing regimen as compared to the standard daily dosing regimen of risedronate 5 mg daily.

DETAILED DESCRIPTION:
The comparator arms of this risedronate study are 150 mg monthly and 5 mg daily.

ELIGIBILITY:
Inclusion Criteria:

* Female: 50 years of age or older
* >5 years since last menses natural or surgical
* have lumbar spine BMD (bone mineral density) more that 2.5 standard deviations (SD) below the young adult mean, or have 1-spine BMD more than 2.0 SD below the young adult female mean value and also have at least one prevalent vertebral body fracture

Exclusion Criteria:

* history of uncontrolled hyperparathyroidism, hyperthyroidism, osteomalacia
* BMI (body mass index) >32 kg/m^2
* use of medications within 3 months of starting study drug that impact bone metabolism such as glucocorticoids, estrogens, calcitonin, calcitriol, other bisphosphonates and parathyroid hormone
* hypocalcemia or hypercalcemia of any cause
* markedly abnormal clinical laboratory measurements that are assessed as clinically significant by the investigator

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1294 (Actual)
Dates: Start 2005-10; Primary Completion 2008-03 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sal Bartelmo, MD, Study Director — P&G
Locations (49):
- United States (7):
  - Research Site, Lakewood, Colorado
  - Research Site, Gainesville, Georgia
  - Research Site, Bethesda, Maryland
  - Research Site, Omaha, Nebraska
  - Research Site, West Haverstraw, New York
  - Research Site, Cincinnati, Ohio
  - Research Site, Portland, Oregon
- Argentina (2):
  - Research Site, Buenos Aires, Buenos Aires
  - Research Site, Capital Federal
- Australia (3):
  - Research Site, Geelong
  - Research Site, Heidelberg, Victoria
  - Research Site, Saint Leonards
- Belgium (5):
  - Research Site, Brussels
  - Research Site, Ghent
  - Research Site, Leuven
  - Research Site, Liège
  - Research Site, Mont Godinne
- Brazil (2):
  - Research Site, Rio de Janeiro
  - Research Site, São Paulo
- Canada (4):
  - Research Site, Calgary
  - Research Site, Montreal
  - Research Site, Sainte-Foy
  - Research Site, Saskatoon
- Estonia (2):
  - Research Site, Pärnu
  - Research Site, Tartu
- Finland (4):
  - Research Site, Helsinki
  - Research Site, Kuopio
  - Research Site, Oulu
  - Research Site, Turku
- France (6):
  - Research Site, Amiens
  - Research Site, Lyon
  - Research Site, Orléans
  - Research Site, Paris
  - Research Site, Toulouse
  - Research Site, Vandœuvre-lès-Nancy
- Hungary (5):
  - Research Site, Balatonfüred
  - Research Site, Budapest
  - Research Site, Győr
  - Research Site, Miskolc
  - Research Site, Nagykanizs
- Research Site, Beirut, Lebanon
- Norway (3):
  - Research Site, Oslo
  - Research Site, Paradis
  - Research Site, Trondheim
- Poland (2):
  - Research Site, Bialystok
  - Research Site, Warsaw
- Spain (3):
  - Research Site, Barcelona
  - Research Site, Granada
  - Research Site, Madrid

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Screening period began 17 Oct '05
Groups:
- 5 mg Risedronate: 5 mg risedronate tablet, once daily for 2 years
- 150 mg Risedronate: 150 mg risedronate taken once a month for 2 years
Period: Overall Study
Arm/Group | 5 mg Risedronate | 150 mg Risedronate
Started | 644 | 650
Intent to Treat Population | 642 (Two subjects not included as they did not take any study medication.) | 650
Completed | 498 | 513
Not Completed | 146 | 137
Not completed — Adverse Event | 85 | 80
Not completed — Physician Decision | 6 | 3
Not completed — Lost to Follow-up | 7 | 7
Not completed — Withdrawal by Subject | 46 | 47
Not completed — Did not take any study drug | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 5 mg Risedronate | 150 mg Risedronate | Total
Number analyzed (Participants) | 644 | 650 | 1294
Age Continuous [Mean (Standard Deviation); unit: years] — ITT (intent to treat) Population
  years | 64.4 (7.7) | 65.5 (7.2) | 64.9 (7.5)
Age, Customized [Number; unit: Partcipants] — ITT Population
  Partcipants
    < 65 years | 335 | 304 | 639
    65 - <75 years | 232 | 268 | 500
    > = 75 years | 75 | 78 | 153
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 644 | 650 | 1294
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — ITT Population
  participants
    Argentina | 302 | 304 | 606
    Australia | 7 | 7 | 14
    Belgium | 13 | 14 | 27
    Canada | 19 | 19 | 38
    Spain | 7 | 9 | 16
    Estonia | 48 | 50 | 98
    Finland | 17 | 18 | 35
    France | 50 | 49 | 99
    Hungary | 22 | 22 | 44
    Lebanon | 6 | 6 | 12
    Norway | 24 | 25 | 49
    Poland | 103 | 104 | 207
    United States | 24 | 23 | 47

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Lumbar Spine Bone Mineral Density (BMD) at Month 12-Endpoint in Women With Postmenopausal Osteoporosis, Primary Efficacy Population
Description: BMD assessed using dual-energy x-ray absorptiometry (DXA) using Hologic or Lunar equipment. LOCF - last observation carried forward (Last post-baseline measurement available to Month 12).
Time Frame: Baseline to Month 12 - Endpoint
Population: ITT (intent to treat) Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | 5 mg Risedronate | 150 mg Risedronate
Number analyzed (Participants) | 642 | 650
Percent Change | 3.425 [3.028 to 3.823] | 3.540 [3.147 to 3.934]
Statistical Analysis 1: Comparison: 5 mg Risedronate vs 150 mg Risedronate; Test type: Non-Inferiority or Equivalence — In order to establish noninferiority for the primary efficacy variable at one-sided α of 2.5% with 90% power, a total of 1068 patients, 534 per treatment group, is required. This calculation is based on the following assumptions: the noninferiority margin (or delta) = 1.5%, the common SD (standard deviation) of the percent change from baseline in lumbar spine BMD at Month 12 = 4.5%, the 1 year dropout rate = 20%, and the true mean difference μD - μM = 0.5%; ANOVA; Fixed effects for treatment and pooled center; Least Square (LS) Mean Difference = -0.115, 95% CI 2-sided [-0.505 to 0.274]

2. Secondary Outcome: Percent Change From Baseline in Lumbar Spine BMD at Month 12, ITT Population
Description: BMD assessed using dual-energy x-ray absorptiometry (DXA) using Hologic or Lunar equipment.
Time Frame: Baseline to Month 12
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | 5 mg Risedronate | 150 mg Risedronate
Number analyzed (Participants) | 642 | 650
Percent Change | 3.522 [3.116 to 3.928] | 3.598 [3.201 to 3.995]
Statistical Analysis 1: Comparison: 5 mg Risedronate vs 150 mg Risedronate; Test type: Superiority or Other; ANOVA; Fixed effects for treatment and pooled center; LS Mean Difference = -0.076, 95% CI 2-sided [-0.475 to 0.323]

3. Secondary Outcome: Change From Baseline in Lumbar Spine BMD at Month 12, ITT Population
Description: BMD assessed using dual-energy x-ray absorptiometry (DXA) using Hologic or Lunar equipment.
Time Frame: Baseline to Month 12
Population: ITT
Measure: Least Squares Mean (95% Confidence Interval); unit: g/cm^2
Arm/Group | 5 mg Risedronate | 150 mg Risedronate
Number analyzed (Participants) | 642 | 650
g/cm^2 | 0.0256 [0.0226 to 0.0286] | 0.0261 [0.0232 to 0.0291]
Statistical Analysis 1: Comparison: 5 mg Risedronate vs 150 mg Risedronate; Test type: Superiority or Other; ANOVA; Fixed effects for treatment and pooled center; LS Mean Difference = -0.0005, 95% CI 2-sided [-0.0035 to 0.0024]

4. Secondary Outcome: Percent Change From Baseline in Lumbar Spine BMD at Month 24-Endpoint, Endpoint Population (Month 24)
Description: BMD assessed using dual-energy x-ray absorptiometry (DXA) using Hologic or Lunar equipment. LOCF - last observation carried forward (Last post-baseline measurement available to Month 24).
Time Frame: Baseline to Month 24 - Endpoint
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | 5 mg Risedronate | 150 mg Risedronate
Number analyzed (Participants) | 642 | 650
Percent Change | 3.927 [3.432 to 4.422] | 4.166 [3.677 to 4.654]
Statistical Analysis 1: Comparison: 5 mg Risedronate vs 150 mg Risedronate; The sample size of 1068 patients will provide approximately 90% power to demonstrate the noninferiority of the monthly regimen at month 24, using a 2% noninferiority margin and assuming a common SD of the percent change from baseline in lumbar spine BMD at month 24 of 5%, a 2-year dropout rate of 30%, and a true mean difference (uDaily-uMonthly) of 0.8%; Test type: Non-Inferiority or Equivalence — The estimates of the common SD, dropout rate at month 24 and true difference are also based on previous risedronate Phase III studies (RVN008993, RVE009093, ROE009394, HMR4003E/3001); ANOVA; Fixed effects for treatment and pooled centers; LS Mean Difference = -0.239, 95% CI 2-sided [-0.727 to 0.249]

5. Secondary Outcome: Percent Change From Baseline in Lumbar Spine BMD at Month 24, ITT Population
Description: BMD assessed using dual-energy x-ray absorptiometry (DXA) using Hologic or Lunar equipment.
Time Frame: Baseline to Month 24
Population: ITT
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | 5 mg Risedronate | 150 mg Risedronate
Number analyzed (Participants) | 642 | 650
Percent Change | 4.217 [3.685 to 4.750] | 4.302 [3.783 to 4.822]
Statistical Analysis 1: Comparison: 5 mg Risedronate vs 150 mg Risedronate; Test type: Superiority or Other; ANOVA; Fixed Effects for treatment & pooled center; Mean Difference (Final Values) = -0.085, 95% CI 2-sided [-0.609 to 0.439]

6. Secondary Outcome: Change From Baseline in Lumbar Spine BMD at Month 24, ITT Population
Description: BMD assessed using dual-energy x-ray absorptiometry (DXA) using Hologic or Lunar equipment.
Time Frame: Baseline to Month 24
Population: ITT
Measure: Least Squares Mean (95% Confidence Interval); unit: g/cm^2
Arm/Group | 5 mg Risedronate | 150 mg Risedronate
Number analyzed (Participants) | 642 | 650
g/cm^2 | 0.0309 [0.0270 to 0.0349] | 0.0319 [0.0280 to 0.0357]
Statistical Analysis 1: Comparison: 5 mg Risedronate vs 150 mg Risedronate; Test type: Superiority or Other; ANOVA; Fixed effects for treatment and pooled center; Mean Difference (Final Values) = -0.0009, 95% CI 2-sided [-0.0048 to 0.0029]

7. Secondary Outcome: Change From Baseline in Urine Type-1 Collagen Cross-linked-N-telopeptide Corrected for Creatinine Clearance (NTX/Cr) at Month 6, ITT Population
Description: Assayed by ELISA (enzyme-linked immunosorbent assay) for NTX and colorimetric assay for creatinine. Patient collected second urine voided between 6 and 9 am from day of clinic visit and day before clinic visit at Months 3, 6, 12 & 24. nmol BCE / mmol Creatinine = nanomoles bone collagen equivalents / millimoles Creatinine
Time Frame: Baseline to Month 6
Population: ITT
Measure: Least Squares Mean (95% Confidence Interval); unit: nmol BCE / mmol Creatinine
Arm/Group | 5 mg Risedronate | 150 mg Risedronate
Number analyzed (Participants) | 642 | 650
nmol BCE / mmol Creatinine | -30.04 [-33.19 to -26.88] | -30.26 [-33.41 to -27.12]
Statistical Analysis 1: Comparison: 5 mg Risedronate vs 150 mg Risedronate; Test type: Superiority or Other; ANOVA; Fixed effects for treatment and pooled center; Mean Difference (Final Values) = 0.23, 95% CI 2-sided [-2.83 to 3.28]

8. Secondary Outcome: Percent Change From Baseline in Urine NTX/Cr at Month 6, ITT Population
Description: Assayed by ELISA (enzyme-linked immunosorbent assay) for NTX and colorimetric assay for creatinine. Patient collected second urine voided between 6 and 9 am from day of clinic visit and day before clinic visit at Months 3, 6, 12 & 24.
Time Frame: Baseline to Month 6
Population: ITT
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | 5 mg Risedronate | 150 mg Risedronate
Number analyzed (Participants) | 642 | 650
Percent Change | -51.83 [-54.83 to -48.83] | -50.26 [-53.25 to -47.27]
Statistical Analysis 1: Comparison: 5 mg Risedronate vs 150 mg Risedronate; Test type: Superiority or Other; ANOVA; Fixed effects for treatment and pooled center; Mean Difference (Final Values) = -1.57, 95% CI 2-sided [-4.47 to 1.33]

9. Secondary Outcome: Change From Baseline in Urine NTX/Cr at Month 24, ITT Population
Description: as for outcome 8
Time Frame: Baseline to Month 24
Population: ITT
Measure: Least Squares Mean (95% Confidence Interval); unit: nmol BCE / mmol Creatinine
Arm/Group | 5 mg Risedronate | 150 mg Risedronate
Number analyzed (Participants) | 642 | 650
nmol BCE / mmol Creatinine | -28.88 [-32.50 to -25.26] | -29.87 [-33.38 to -26.37]
Statistical Analysis 1: Comparison: 5 mg Risedronate vs 150 mg Risedronate; Test type: Superiority or Other; ANOVA; Fixed effects for treatment and pooled center; Mean Difference (Final Values) = 1.00, 95% CI 2-sided [-2.54 to 4.53]

10. Secondary Outcome: Percent Change From Baseline in Urine NTX/Cr at Month 24, ITT Population
Description: as for outcome 8
Time Frame: Baseline to Month 24
Population: ITT
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | 5 mg Risedronate | 150 mg Risedronate
Number analyzed (Participants) | 642 | 650
Percent Change | -49.45 [-53.16 to -45.74] | -46.62 [-50.21 to -43.03]
Statistical Analysis 1: Comparison: 5 mg Risedronate vs 150 mg Risedronate; Test type: Superiority or Other; ANOVA; Fixed effects for treatment and pooled center; Mean Difference (Final Values) = -2.83, 95% CI 2-sided [-6.45 to 0.80]

11. Secondary Outcome: Change From Baseline in Serum Type-1 Collagen Cross-linked C-telopeptide (CTX) at Month 6, ITT Population
Description: ng / mL = nanograms / milliliter. Assayed by electrochemiluminescent immunoassay.
Time Frame: Baseline to Month 6
Population: ITT
Measure: Least Squares Mean (95% Confidence Interval); unit: ng / mL
Arm/Group | 5 mg Risedronate | 150 mg Risedronate
Number analyzed (Participants) | 642 | 650
ng / mL | -0.36 [-0.39 to -0.33] | -0.34 [-0.37 to -0.31]
Statistical Analysis 1: Comparison: 5 mg Risedronate vs 150 mg Risedronate; Test type: Superiority or Other; ANOVA; Fixed effects for treatment and pooled center; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.05 to 0.00]

12. Secondary Outcome: Percent Change From Baseline in Serum CTX at Month 6, ITT Population
Description: Assayed by electrochemiluminescent immunoassay.
Time Frame: Baseline to Month 6
Population: ITT
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | 5 mg Risedronate | 150 mg Risedronate
Number analyzed (Participants) | 642 | 650
Percent Change | -57.79 [-61.73 to -53.84] | -53.62 [-57.54 to -49.69]
Statistical Analysis 1: Comparison: 5 mg Risedronate vs 150 mg Risedronate; Test type: Superiority or Other; ANOVA; Fixed effects for treatment and pooled center; Mean Difference (Final Values) = -4.17, 95% CI 2-sided [-7.98 to -0.36]

13. Secondary Outcome: Change From Baseline in Serum CTX at Month 24, ITT Population
Description: Assayed by electrochemiluminescent immunoassay.
Time Frame: Baseline to Month 24
Population: ITT
Measure: Least Squares Mean (95% Confidence Interval); unit: ng / mL
Arm/Group | 5 mg Risedronate | 150 mg Risedronate
Number analyzed (Participants) | 642 | 650
ng / mL | -0.22 [-0.26 to -0.19] | -0.20 [-0.23 to -0.17]
Statistical Analysis 1: Comparison: 5 mg Risedronate vs 150 mg Risedronate; Test type: Superiority or Other; ANOVA; Fixed effects for treatment and pooled center; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.06 to 0.01]

14. Secondary Outcome: Percent Change From Baseline in Serum CTX at Month 24, ITT Population
Description: Assayed by electrochemiluminescent immunoassay.
Time Frame: Baseline to Month 24
Population: ITT
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | 5 mg Risedronate | 150 mg Risedronate
Number analyzed (Participants) | 642 | 650
Percent Change | -29.33 [-35.82 to -22.84] | -23.63 [-29.94 to -17.33]
Statistical Analysis 1: Comparison: 5 mg Risedronate vs 150 mg Risedronate; Test type: Superiority or Other; ANOVA; Fixed effects for treatment and pooled center; Mean Difference (Final Values) = -5.69, 95% CI 2-sided [-12.04 to 0.66]

15. Secondary Outcome: Change From Baseline in Serum Bone-specific Alkaline Phosphatase (BAP) at Month 6, ITT Population
Description: ug / L = micrograms per liter, Assayed by ELISA (enzyme-linked immunosorbent assay)
Time Frame: Baseline to Month 6
Population: ITT
Measure: Least Squares Mean (95% Confidence Interval); unit: ug / L
Arm/Group | 5 mg Risedronate | 150 mg Risedronate
Number analyzed (Participants) | 642 | 650
ug / L | -5.31 [-5.79 to -4.83] | -5.48 [-5.96 to -5.00]
Statistical Analysis 1: Comparison: 5 mg Risedronate vs 150 mg Risedronate; Test type: Superiority or Other; ANOVA; Fixed effects for treatment and pooled center; Mean Difference (Final Values) = 0.17, 95% CI 2-sided [-0.29 to 0.64]

16. Secondary Outcome: Percent Change From Baseline in Serum BAP at Month 6, ITT Population
Description: Assayed by ELISA (enzyme-linked immunosorbent assay)
Time Frame: Baseline to Month 6
Population: ITT
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | 5 mg Risedronate | 150 mg Risedronate
Number analyzed (Participants) | 642 | 650
Percent Change | -33.34 [-35.58 to -31.11] | -34.66 [-36.88 to -32.43]
Statistical Analysis 1: Comparison: 5 mg Risedronate vs 150 mg Risedronate; Test type: Superiority or Other; ANOVA; Fixed effects for treatment and pooled center; Mean Difference (Final Values) = 1.31, 95% CI 2-sided [-0.85 to 3.48]

17. Secondary Outcome: Change From Baseline in Serum BAP at Month 24, ITT Population
Description: Assayed by ELISA (enzyme-linked immunosorbent assay)
Time Frame: Baseline to Month 24
Population: ITT
Measure: Least Squares Mean (95% Confidence Interval); unit: ug / L
Arm/Group | 5 mg Risedronate | 150 mg Risedronate
Number analyzed (Participants) | 642 | 650
ug / L | -4.10 [-4.69 to -3.52] | -4.22 [-4.79 to -3.65]
Statistical Analysis 1: Comparison: 5 mg Risedronate vs 150 mg Risedronate; Test type: Superiority or Other; ANOVA; Fixed effects for treatment and pooled center; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [-0.45 to 0.70]

18. Secondary Outcome: Percent Change From Baseline in Serum BAP at Month 24, ITT Population
Description: Assayed by ELISA (enzyme-linked immunosorbent assay)
Time Frame: Baseline to Month 24
Population: ITT
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | 5 mg Risedronate | 150 mg Risedronate
Number analyzed (Participants) | 642 | 650
Percent Change | -25.84 [-29.10 to -22.57] | -25.07 [-28.25 to -21.90]
Statistical Analysis 1: Comparison: 5 mg Risedronate vs 150 mg Risedronate; Test type: Superiority or Other; ANOVA; Fixed effects for treatment and pooled center; Mean Difference (Final Values) = -0.77, 95% CI 2-sided [-3.96 to 2.43]

19. Secondary Outcome: Number of Participants With New Vertebral Fracture at Month 12, ITT Population
Description: At least 1 new fractured vertebra
Time Frame: Baseline to Month 12
Population: ITT
Measure: Number; unit: Participants
Arm/Group | 5 mg Risedronate | 150 mg Risedronate
Number analyzed (Participants) | 642 | 650
Participants | 8 | 8
Statistical Analysis 1: Comparison: 5 mg Risedronate vs 150 mg Risedronate; Test type: Superiority or Other; p = 1.0000, Fisher Exact; Risk Ratio (RR) = 0.96, 95% CI 2-sided [0.36 to 2.54]

20. Secondary Outcome: Number of Participants With New Vertebral Fracture at Month 24, ITT Population
Description: At least 1 new fractured vertebra
Time Frame: Baseline to Month 24
Population: ITT
Measure: Number; unit: Participants
Arm/Group | 5 mg Risedronate | 150 mg Risedronate
Number analyzed (Participants) | 642 | 650
Participants | 14 | 14
Statistical Analysis 1: Comparison: 5 mg Risedronate vs 150 mg Risedronate; Test type: Superiority or Other; p = 1.0000, Fisher Exact; Risk Ratio (RR) = 0.98, 95% CI 2-sided [0.47 to 2.03]

ADVERSE EVENTS:
Time Frame: 17 Oct '05 thru 18 Mar '08
Arm/Group | 5 mg Risedronate | 150 mg Risedronate
Serious Adverse Events (participants affected / at risk) | 51/642 | 77/650
Other Adverse Events (participants affected / at risk) | 554/642 | 578/650
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5 mg Risedronate (N=642) | 150 mg Risedronate (N=650)
Myocardial Ischaemia (Cardiac disorders) | 1 (1) | 3 (3)
Acute Coronary Syndrome (Cardiac disorders) | 0 (0) | 2 (3)
Angina Unstable (Cardiac disorders) | 0 (0) | 2 (2)
Angina Pectoris (Cardiac disorders) | 1 (1) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 3 (4)
Congestive Cardiomyopathy (Cardiac disorders) | 1 (1) | 1 (1)
Hypertrophic Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 1 (1) | 1 (1)
Aortic Valve Incompetence (Cardiac disorders) | 1 (2) | 0 (0)
Cardiac Failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 2 (2) | 3 (3)
Ischaemic Stroke (Nervous system disorders) | 0 (0) | 1 (1)
Carotid Artery Stenosis (Nervous system disorders) | 0 (0) | 1 (1)
Vertebrobasilar Insufficiency (Nervous system disorders) | 0 (0) | 1 (1)
Loss of Consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Transient Ischaemic Attack (Nervous system disorders) | 0 (0) | 2 (2)
Dementia Alzheimer's Type (Nervous system disorders) | 0 (0) | 1 (1)
Facial Palsy (Nervous system disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
Lumbar Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Cubital Tunnel Syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Parkinson's Disease (Nervous system disorders) | 1 (1) | 0 (0)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 7 (7)
Benign Neoplasm of Thyroid Gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thyroid Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Fibroadenoma of Breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebellar Tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung Adenocarcinoma Stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colorectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Parathyroid Tumour Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Acute Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to Lymph Nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal Cell Carcinoma Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Bronchopneumonia (Infections and infestations) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 5 (6) | 2 (2)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 2 (2)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Postoperative Abscess (Infections and infestations) | 0 (0) | 1 (1)
Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Toxoplasmosis (Infections and infestations) | 0 (0) | 1 (1)
Chronic Sinusitis (Infections and infestations) | 0 (0) | 1 (2)
Pharyngolaryngeal abscess (Infections and infestations) | 1 (1) | 0 (0)
Filariasis (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Lymphangitis (Infections and infestations) | 1 (1) | 0 (0)
Patella Fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Femur Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fibula Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tibia Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip Fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Hand Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Humerus Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radius Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wrist Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pancreatitis Acute (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 1 (1)
Erosive Duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Adbominal Pain Upper (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Intestinal Prolapse (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis Erosive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Subileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large Intestine Perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Umbilical Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cholelithiasis (Gastrointestinal disorders) | 2 (2) | 4 (4)
Hepatic Cyst (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cholangitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bile Duct Stone (Gastrointestinal disorders) | 0 (0) | 1 (1)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Eosinophilic Fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Foot Deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Vaginal Prolapse (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Colpocele (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Rectocele (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Cystocele (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cervical Dysplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 3 (3)
Asthmatic Crisis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypertensive Emergency (Vascular disorders) | 0 (0) | 1 (1)
Aortic Dilatation (Vascular disorders) | 0 (0) | 1 (1)
Varicose Vein (Vascular disorders) | 1 (1) | 1 (1)
Cardiovascular Insufficiency (Vascular disorders) | 1 (1) | 0 (0)
Bladder Prolapse (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urethral Stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Calculus Urinary (Renal and urinary disorders) | 1 (1) | 0 (0)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Chest Pain (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Major Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Blindness (Eye disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Drug Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pemphigoid (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Drug Eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5 mg Risedronate (N=642) | 150 mg Risedronate (N=650)
Influenza (Infections and infestations) | 57 (62) | 94 (112)
Nasopharyngitis (Infections and infestations) | 62 (76) | 70 (86)
Urinary Tract Infection (Infections and infestations) | 50 (58) | 61 (83)
Bronchitis (Infections and infestations) | 68 (76) | 57 (74)
Diarrrhoea (Gastrointestinal disorders) | 43 (49) | 69 (95)
Abdominal Pain Upper (Gastrointestinal disorders) | 51 (65) | 62 (74)
Nausea (Gastrointestinal disorders) | 52 (61) | 47 (56)
Dyspepsia (Gastrointestinal disorders) | 37 (41) | 44 (52)
Constipation (Gastrointestinal disorders) | 53 (56) | 43 (52)
Vomiting (Gastrointestinal disorders) | 32 (36) | 36 (41)
Arthralgia (Musculoskeletal and connective tissue disorders) | 68 (81) | 65 (76)
Back Pain (Musculoskeletal and connective tissue disorders) | 80 (87) | 65 (73)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 35 (37) | 45 (50)
Headache (Nervous system disorders) | 38 (51) | 35 (37)
Fall (Injury, poisoning and procedural complications) | 45 (57) | 57 (66)
Hypertension (Vascular disorders) | 49 (53) | 52 (55)
Gastroenteritis (Infections and infestations) | 21 (24) | 24 (25)
Upper Respiratory Tract Infection (Infections and infestations) | 11 (12) | 18 (24)
Pneumonia (Infections and infestations) | 7 (10) | 13 (13)
Tooth Infection (Infections and infestations) | 13 (14) | 11 (16)
Cystitis (Infections and infestations) | 19 (22) | 10 (11)
Sinusitis (Infections and infestations) | 15 (15) | 10 (10)
Pharyngitis (Infections and infestations) | 14 (15) | 9 (10)
Abdominal Pain (Gastrointestinal disorders) | 32 (36) | 31 (48)
Gastritis (Gastrointestinal disorders) | 19 (21) | 24 (26)
Abdominal Distention (Gastrointestinal disorders) | 16 (18) | 19 (24)
Flatulence (Gastrointestinal disorders) | 19 (19) | 18 (21)
Hyperchlorhydria (Gastrointestinal disorders) | 4 (4) | 18 (18)
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 13 (14) | 11 (11)
Hiatus Hernia (Gastrointestinal disorders) | 20 (20) | 8 (8)
Gastritis erosive (Gastrointestinal disorders) | 14 (15) | 7 (7)
Dry Mouth (Gastrointestinal disorders) | 13 (13) | 3 (3)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 24 (28) | 29 (31)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 14 (15) | 22 (23)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 20 (21) | 20 (22)
Myalgia (Musculoskeletal and connective tissue disorders) | 12 (13) | 17 (19)
Tendonitis (Musculoskeletal and connective tissue disorders) | 16 (17) | 16 (16)
Neck Pain (Musculoskeletal and connective tissue disorders) | 19 (20) | 15 (15)
Muscle Contracture (Musculoskeletal and connective tissue disorders) | 14 (14) | 6 (6)
Dizziness (Nervous system disorders) | 17 (20) | 26 (27)
Sciatica (Nervous system disorders) | 11 (12) | 17 (19)
Contusion (Injury, poisoning and procedural complications) | 19 (26) | 17 (24)
Asthenia (General disorders) | 18 (19) | 23 (24)
Chest Pain (General disorders) | 11 (11) | 21 (21)
Oedema Peripheral (General disorders) | 10 (11) | 14 (14)
Pyrexia (General disorders) | 8 (9) | 13 (25)
Cough (Respiratory, thoracic and mediastinal disorders) | 20 (22) | 24 (25)
Alopecia (Skin and subcutaneous tissue disorders) | 7 (7) | 14 (16)
Pruritus (Skin and subcutaneous tissue disorders) | 19 (22) | 10 (14)
Depression (Psychiatric disorders) | 19 (19) | 20 (21)
Anxiety (Psychiatric disorders) | 13 (13) | 18 (18)
Insomnia (Psychiatric disorders) | 16 (16) | 9 (9)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 12 (12) | 22 (22)
Cataract (Eye disorders) | 12 (13) | 16 (19)
Conjunctivitis (Eye disorders) | 6 (6) | 13 (13)
Vertigo (Ear and labyrinth disorders) | 9 (11) | 17 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less